CLINICAL TRIAL: NCT01955031
Title: Effectiveness and Cost-effectiveness Analysis of a Telemonitoring Program on Lifestyle for People With Type 2 Diabetes at Home. Study Based on a Health Network in Diabetology.
Brief Title: Effectiveness and Cost-effectiveness of a Telemonitoring Program for Diabetic People at Home
Acronym: EDUC@DOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12 424 03; PREPS (Other: CHU de Toulouse)
Record Dates: First submitted 2013-08-22; First posted 2013-10-07 (Estimated); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Type 2 Diabetes
Keywords: Telemedicine; Telemonitoring; Education; Nutrition; Food behaviour; Weight; Physical activity; Glycaemia; Self-monitoring blood glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Body Weight; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telemonitoring (Experimental): Patient with type 2 diabetes randomized in telemonitoring group have a telemonitoring device with educational Tools at their home
  Interventions: Other: telemonitoring
- Usual care (Sham Comparator): patient randomized in this group have a usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Other: telemonitoring — A telemonitoring program with educational tools is given to people with type 2 diabetes at their home. It is composed of three softwares to improve eating habits available on touchpad, a self-monitoring blood glucose device, a balance to measure weight and fat mass, and a pedometer to evaluate physical activity. Data are securely sent and stored into a web service which delivers a synthesis to patients and health professionals.
  Arms: Telemonitoring
Other: Usual care — Patients are recruited during therapeutic educational sessions or appointments by general practitioners or diabetologists who take part into the Regional Health Network in Diabetes DIAMIP. If patients accept to participate to the study and sign up the protocol consent, they are given questionnaires about nutrition, physical activity and quality of life. A dietician analyses with each patient the results of a food inquiry. Patients are randomised into two groups: one arm is trained to the telemonitoring program before receiving it at home, and the other arm follows usual care. During 12 months, the telemonitoring group uses the device. The investigators (GP or diabetologists) can use the specific secured website to follow the measured parameters and to make appropriate decisions about health care of their patient. No consultation are scheduled in advance.
  Arms: Usual care

SUMMARY:
Severity of diabetes is related to the development of disabling and costly complications (12.9 billion euros in 2007). The French High Health Authority recommends a therapeutic education on lifestyle and dietary rules in first-line treatment of Type 2 Diabetes Mellitus. Despite these recommendations, patients often have difficulties to implement dietary recommendations every day. The objective of EDUC@DOM is to help people with diabetes to improve lifestyle and equilibrium of glycaemia in order to avoid or delay chronic complications of diabetes. Our main goal is to assess effectiveness of our telemonitoring program in type 2 patients' care compared to a usual care of diabetes, on the glycaemia of the patients. It is expected that our program leads to a better monitoring of health status, a greater adherence to medical and non-medical prescriptions, an empowerment of the patient, and as a consequence, a more efficient health care consumption.

ELIGIBILITY:
Inclusion Criteria:

* Patient with type 2 diabetes
* Older than 18 years
* With an insulin treatment or not
* Having a glycemic impairment characterized by 6.5% <HbA1c ≤10
* Having an active internet connection at home.
* Accepting the terms of training, loan and use of the device
* Benefiting from social protection system
* Having given his/her free and informed consent and signed the consent

Exclusion Criteria:

* Serious illness recently (<3 months) or decompensated may influence glycemic control of the patient permanently according to the judgment of the physician in charge of monitoring
* Retinal state that does not allow optimization in equilibrium of glycaemia
* Known severe renal impairment defined by creatinine clearance <30ml/min
* Known hemoglobinopathy
* Visual or intellectual resulting inability to use the remote monitoring tool according to the judgment of the physician in charge of monitoring
* Inability to understand all or part of the software information according to the judgment of the physician in charge of monitoring
* Subject to disabled
* Person with severe behavioral disorders (anorexia, bulimia, ...) according to the judgment of the physician in charge of monitoring
* Person who had, or in preparation for bariatric surgery (software nutrition education are not suitable for this type of care.)
* Person with a medical device implanted electronic pacemakers and defibrillators with cardiac (possibility of interference with the impedance)
* Another person involved in research including a period of ongoing exclusion to inclusion,
* A person under legal protection
* Subject living in institutions
* Desire for pregnancy, pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2013-11; Primary Completion 2016-05 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
To assess effectiveness of our telemonitoring program in Diabetes care, HbA1C assays will be compared between the two groups.The change of HbA1c between day 0, month 1,month 3, month 6, month 9 and month 12 | HbA1c will be measured at Day 0, month 1, month 3, month 6, month 9 and month 12

SECONDARY OUTCOMES:
Assessment efficacy of our program by the measure of HbA1C will | At month 15, month 18, month 21 and month 24
Questionnaires will be given to patients to assess the improvement of nutritional knowledge | At day 0 and month 24
Food inquiries will be given to patients to assess the improvement of eating habits | At day 0 and month 24
Questionnaires will be given to patients to assess the physical activity practice | At day 0 and month 24
Waist circumference will be measured to assess the body composition, BMI (Body Mass Index), | At day 0 and month 24
The self-monitoring blood glucose books will be copied to assess mean of blood glycaemia | At day 0, month 12 and month 24
A blood sample will be collected to assess lipid status | At day 0 and month 24
Two questionnaires will be given to patients to assess quality of life of patients | At day 0 and month 24
A cost-effectiveness ratio and a markov modelisation will be realized to assess the economic aspects | At month 24
For the telemonitoring arm, assessment of food behavior through meals registered with the Nutri-Educ software | Everytime patients use the software from Day 0 to month 24
For the telemonitoring arm, assessment of nutritional knowledge through rate of good choices playing games of Nutri-Kiosk software | Everytime patients use the software from Day0 to month 24
For the telemonitoring arm, assessment of physical activity declared through Acti-Kiosk software and measures collected with the pedometer (number of steps, number of stairs climbed up) | Every time patients use the software and the pedometer from day 0 to month 24
For the telemonitoring arm, measure of weight, fat rate and lean rate collected with the balance | Everytime patients use the balance from day 0 to month 24
For the telemonitoring arm, means of glycaemia collected with the self-monitoring blood glucose device | Everytime patients use the blood glucose device from day 0 to month 24
For the telemonitoring arm, acceptability and satisfaction of the telemonitoring system by the patients with the number and time of connections and a questionnaire | At month 24
For the telemonitoring arm, acceptability and satisfaction of the telemonitoring system by the health professionals with the number and time of connections | At month 24
For the telemonitoring arm, acceptability and satisfaction of the telemonitoring system by the health professionals with the number and time of connections leading to a medical decision (phone call or medical appointment) and a questionnaire | At month 24

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Christine TURNIN, MD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University Hospitals of Toulouse (Rangueil and Salies-Du-Salat), Toulouse, Midi-Pyrénées, France

REFERENCES:
- [Background] InVS (Institut de veille sanitaire). Fagot-Campagna Anne, Romon Isabelle, Fosse Sandrine, Roudier Candice. Prévalence et incidence du diabète, et mortalité liée au diabète en France Synthèse épidémiologique. Novembre 2010
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] HAS (Haute Autorité de Santé). Agence Nationale de sécurité du médicament et des produits de santé. Recommandations de bonne pratique. Stratégie médicamenteuse du contrôle glycémique du diabète de type 2. Janvier 2013.
- [Background] HAS (Haute Autorité de Santé). Rapport d'orientation - Développement de la prescription de thérapeutiques non médicamenteuses validées - Avril 2011
- [Background] Trento M, Gamba S, Gentile L, Grassi G, Miselli V, Morone G, Passera P, Tonutti L, Tomalino M, Bondonio P, Cavallo F, Porta M; ROMEO Investigators. Rethink Organization to iMprove Education and Outcomes (ROMEO): a multicenter randomized trial of lifestyle intervention by group care to manage type 2 diabetes. Diabetes Care. 2010 Apr;33(4):745-7. doi: 10.2337/dc09-2024. Epub 2010 Jan 26. PMID 20103547
- [Background] Welschen LM, Bloemendal E, Nijpels G, Dekker JM, Heine RJ, Stalman WA, Bouter LM. Self-monitoring of blood glucose in patients with type 2 diabetes who are not using insulin: a systematic review. Diabetes Care. 2005 Jun;28(6):1510-7. doi: 10.2337/diacare.28.6.1510. No abstract available. PMID 15920083
- [Background] Norris SL, Engelgau MM, Narayan KM. Effectiveness of self-management training in type 2 diabetes: a systematic review of randomized controlled trials. Diabetes Care. 2001 Mar;24(3):561-87. doi: 10.2337/diacare.24.3.561. PMID 11289485
- [Background] INPES (Institut National de Prévention et d'Education pour la Santé). Labalette Céline, Buttet Pierre, Marchand Annie-Claude - DDESET. L'éducation thérapeutique du patient dans les schémas régionaux d'organisation sanitaire de 3e génération 2006-2011. Education thérapeutique du patient dans les Sros 3-INPES- 2007
- [Background] HAS (Haute Autorité de Santé) et INPES (Institut National de Prévention et d'Education pour la Santé). Guide Méthodologique. Structuration d'un programme d'éducation thérapeutique du patient dans le champ des maladies chroniques. Juin 2007
- [Background] MINISTÈRE DE LA SANTÉ ET DES SPORTS - Décret no 2010-904 du 2 août 2010 relatif aux conditions d'autorisation des programmes d'éducation thérapeutique du patient, - Décret no 2010-906 du 2 août 2010 relatif aux compétences requises pour dispenser l'éducation thérapeutique du patient - Arrêté du 2 août 2010 relatif aux compétences requises pour dispenser l'éducation thérapeutique du patient - Arrêté du 2 août 2010 relatif au cahier des charges des programmes d'éducation thérapeutique du patient et à la composition du dossier de demande de leur autorisation
- [Background] Polisena J, Tran K, Cimon K, Hutton B, McGill S, Palmer K. Home telehealth for diabetes management: a systematic review and meta-analysis. Diabetes Obes Metab. 2009 Oct;11(10):913-30. doi: 10.1111/j.1463-1326.2009.01057.x. Epub 2009 Jun 16. PMID 19531058
- [Background] McMahon GT, Gomes HE, Hickson Hohne S, Hu TM, Levine BA, Conlin PR. Web-based care management in patients with poorly controlled diabetes. Diabetes Care. 2005 Jul;28(7):1624-9. doi: 10.2337/diacare.28.7.1624. PMID 15983311
- [Background] Quinn CC, Clough SS, Minor JM, Lender D, Okafor MC, Gruber-Baldini A. WellDoc mobile diabetes management randomized controlled trial: change in clinical and behavioral outcomes and patient and physician satisfaction. Diabetes Technol Ther. 2008 Jun;10(3):160-8. doi: 10.1089/dia.2008.0283. PMID 18473689
- [Background] Shea S, Weinstock RS, Teresi JA, Palmas W, Starren J, Cimino JJ, Lai AM, Field L, Morin PC, Goland R, Izquierdo RE, Ebner S, Silver S, Petkova E, Kong J, Eimicke JP; IDEATel Consortium. A randomized trial comparing telemedicine case management with usual care in older, ethnically diverse, medically underserved patients with diabetes mellitus: 5 year results of the IDEATel study. J Am Med Inform Assoc. 2009 Jul-Aug;16(4):446-56. doi: 10.1197/jamia.M3157. Epub 2009 Apr 23. PMID 19390093
- [Background] Young RJ, Taylor J, Friede T, Hollis S, Mason JM, Lee P, Burns E, Long AF, Gambling T, New JP, Gibson JM. Pro-active call center treatment support (PACCTS) to improve glucose control in type 2 diabetes: a randomized controlled trial. Diabetes Care. 2005 Feb;28(2):278-82. doi: 10.2337/diacare.28.2.278. PMID 15677779
- [Background] Franc S., Dardari D., Boucherie B., Daoudi A., Charpentier G. La télémédecine appliquée au diabète : les résultats acquis et les perspectives à venir. Médecine des maladies Métaboliques, Vol 4, No 3, 2010.
- [Background] Kroeze W, Werkman A, Brug J. A systematic review of randomized trials on the effectiveness of computer-tailored education on physical activity and dietary behaviors. Ann Behav Med. 2006 Jun;31(3):205-23. doi: 10.1207/s15324796abm3103_2. PMID 16700634
- [Background] Brug J, Oenema A, Kroeze W, Raat H. The internet and nutrition education: challenges and opportunities. Eur J Clin Nutr. 2005 Aug;59 Suppl 1:S130-7; discussion S138-9. doi: 10.1038/sj.ejcn.1602186. PMID 16052181
- [Background] Paré Guy, Moqadem Khalil, Pineau Gilles, St-Hilaire Carole. Revue systématique des effets de la télésurveillance à domicile dans le contexte du diabète, des maladies pulmonaires et des maladies cardiovasculaires. AGENCE D'ÉVALUATION DES TECHNOLOGIES ET DES MODES D'INTERVENTION EN SANTÉ. Québec. ETMIS 2009; VOL. 5 : NO 3.
- [Background] Guide Affection de Longue Durée (ALD 8) - Diabète de type 2 - Guide Médecin - juillet 2007
- [Background] Buisson JC. Nutri-Educ, a nutrition software application for balancing meals, using fuzzy arithmetic and heuristic search algorithms. Artif Intell Med. 2008 Mar;42(3):213-27. doi: 10.1016/j.artmed.2007.12.001. Epub 2008 Feb 7. PMID 18261889
- [Background] Buisson J.-C., Garel A. Balancing Meals Using Fuzzy Arithmetics and Heuristic Search Algorithms. IEEE Transactions on Fuzzy Systems, IEEE, Vol. 11 N. 1, p. 68-78, 2003.
- [Background] Turnin MC, Bourgeois O, Cathelineau G, Leguerrier AM, Halimi S, Sandre-Banon D, Coliche V, Breux M, Verlet E, Labrousse F, Bensoussan D, Grenier JL, Poncet MF, Tordjmann F, Brun JM, Blickle JF, Mattei C, Bolzonella C, Buisson JC, Fabre D, Tauber JP, Hanaire-Broutin H. Multicenter randomized evaluation of a nutritional education software in obese patients. Diabetes Metab. 2001 Apr;27(2 Pt 1):139-47. PMID 11353880
- [Background] American Diabetes Association. Standards of medical care in diabetes--2010. Diabetes Care. 2010 Jan;33 Suppl 1(Suppl 1):S11-61. doi: 10.2337/dc10-S011. No abstract available. PMID 20042772
- [Background] Turnin MC, Bolzonella-Pene C, Dumoulin S, Cerf I, Charpentier G, Sandre-Banon D, Valensi P, Grenier JL, Cathelineau G, Mattei C, et al. [Multicenter evaluation of the Nutri-Expert Telematic System in diabetic patients]. Diabete Metab. 1995 Feb;21(1):26-33. French. PMID 7781839
- [Background] Turnin MC, Beddok RH, Clottes JP, Martini PF, Abadie RG, Buisson JC, Soule-Dupuy C, Bonneu M, Camare R, Anton JP, et al. Telematic expert system Diabeto. New tool for diet self-monitoring for diabetic patients. Diabetes Care. 1992 Feb;15(2):204-12. doi: 10.2337/diacare.15.2.204. PMID 1547677
- [Background] Couillard C, Despres JP, Lamarche B, Bergeron J, Gagnon J, Leon AS, Rao DC, Skinner JS, Wilmore JH, Bouchard C. Effects of endurance exercise training on plasma HDL cholesterol levels depend on levels of triglycerides: evidence from men of the Health, Risk Factors, Exercise Training and Genetics (HERITAGE) Family Study. Arterioscler Thromb Vasc Biol. 2001 Jul;21(7):1226-32. doi: 10.1161/hq0701.092137. PMID 11451756
- [Background] Haute Autorité de Santé. BON USAGE DES TECHNOLOGIES DE SANTÉ. L'autosurveillance glycémique dans le diabète de type 2 : une utilisation très ciblée. Avril 2011
- [Background] MINISTÈRE DU TRAVAIL, DE L'EMPLOI ET DE LA SANTÉ. Arrêté du 25 février 2011 relatif à la modification des conditions de prise en charge des appareils pour lecture automatique de la glycémie, dits lecteurs de glycémie, inscrits au chapitre 1er du titre Ier de la liste des produits et prestations remboursables prévue à l'article L. 165-1 du code de la sécurité sociale. JOURNAL OFFICIEL DE LA RÉPUBLIQUE FRANÇAISE. 27 février 2011
- [Background] Jeppsson JO, Kobold U, Barr J, Finke A, Hoelzel W, Hoshino T, Miedema K, Mosca A, Mauri P, Paroni R, Thienpont L, Umemoto M, Weykamp C; International Federation of Clinical Chemistry and Laboratory Medicine (IFCC). Approved IFCC reference method for the measurement of HbA1c in human blood. Clin Chem Lab Med. 2002 Jan;40(1):78-89. doi: 10.1515/CCLM.2002.016. PMID 11916276
- [Background] Hoelzel W, Weykamp C, Jeppsson JO, Miedema K, Barr JR, Goodall I, Hoshino T, John WG, Kobold U, Little R, Mosca A, Mauri P, Paroni R, Susanto F, Takei I, Thienpont L, Umemoto M, Wiedmeyer HM; IFCC Working Group on HbA1c Standardization. IFCC reference system for measurement of hemoglobin A1c in human blood and the national standardization schemes in the United States, Japan, and Sweden: a method-comparison study. Clin Chem. 2004 Jan;50(1):166-74. doi: 10.1373/clinchem.2003.024802. PMID 14709644
- [Background] Weykamp C, John WG, Mosca A, Hoshino T, Little R, Jeppsson JO, Goodall I, Miedema K, Myers G, Reinauer H, Sacks DB, Slingerland R, Siebelder C. The IFCC Reference Measurement System for HbA1c: a 6-year progress report. Clin Chem. 2008 Feb;54(2):240-8. doi: 10.1373/clinchem.2007.097402. PMID 18223132
- [Background] Consensus Committee. Consensus statement on the worldwide standardization of the hemoglobin A1C measurement: the American Diabetes Association, European Association for the Study of Diabetes, International Federation of Clinical Chemistry and Laboratory Medicine, and the International Diabetes Federation. Diabetes Care. 2007 Sep;30(9):2399-400. doi: 10.2337/dc07-9925. No abstract available. PMID 17726190
- [Background] AFSSAPS. Direction de l'Evaluation des Dispositifs Médicaux, Département Surveillance du Marché, Unité Evaluation et Contrôle du Marché - DIV, Dossier suivi par Françoise Chevenne. CAHIER DES CHARGES RELATIF AUX NOTICES DES REACTIFS DOSANT L'HbA1c. Version du 10 janvier 2006
- [Background] Agence Française de Sécurité Sanitaire des Aliments (AFSSA). Avis de l'Agence française de sécurité sanitaire des aliments relatif à l'actualisation des apports nutritionnels conseillés pour les acides gras. Saisine n° 2006-SA-0359. Mars 2010
- [Background] ALFEDIAM PARAMEDICAL Recommandations de Bonnes pratiques. Alimentation du diabétique de type 2. Juin 2003
- [Background] Gautier JF. [Physical activity and type 2 diabetes]. Rev Med Liege. 2005 May-Jun;60(5-6):395-401. French. PMID 16035300
- [Background] GAUTIER JF et al. ACTIVITE PHYSIQUE ET DIABETE 1998 Recommandations de l'Alfediam. Diabetes & metabolism1998, 24:281-290
- [Background] HAS Traitement médicamenteux du diabète de type 2 (actualisation). Novembre 2006.
- [Background] American Diabetes Association. Physical activity/exercise and diabetes. Diabetes Care. 2004 Jan;27 Suppl 1:S58-62. doi: 10.2337/diacare.27.2007.s58. No abstract available. PMID 14693927
- [Background] Sigal RJ, Kenny GP, Wasserman DH, Castaneda-Sceppa C, White RD. Physical activity/exercise and type 2 diabetes: a consensus statement from the American Diabetes Association. Diabetes Care. 2006 Jun;29(6):1433-8. doi: 10.2337/dc06-9910. No abstract available. PMID 16732040
- [Background] Parmenter K, Wardle J. Development of a general nutrition knowledge questionnaire for adults. Eur J Clin Nutr. 1999 Apr;53(4):298-308. doi: 10.1038/sj.ejcn.1600726. PMID 10334656
- [Background] Bongard V, Ruidavets JB, Dallongeville J, Simon C, Amouyel P, Arveiler D, Ducimetiere P, Ferrieres J. Nutritional intakes of 1072 French free-living men with and without diagnosed cardiovascular risk factors. Eur J Clin Nutr. 2004 May;58(5):787-95. doi: 10.1038/sj.ejcn.1601878. PMID 15116082
- [Background] Bull FC, Maslin TS, Armstrong T. Global physical activity questionnaire (GPAQ): nine country reliability and validity study. J Phys Act Health. 2009 Nov;6(6):790-804. doi: 10.1123/jpah.6.6.790. PMID 20101923
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Reliability and validity of a diabetes quality-of-life measure for the diabetes control and complications trial (DCCT). The DCCT Research Group. Diabetes Care. 1988 Oct;11(9):725-32. doi: 10.2337/diacare.11.9.725. PMID 3066604
- [Background] Montori VM, Dinneen SF, Gorman CA, Zimmerman BR, Rizza RA, Bjornsen SS, Green EM, Bryant SC, Smith SA; Translation Project Investigator Group. The impact of planned care and a diabetes electronic management system on community-based diabetes care: the Mayo Health System Diabetes Translation Project. Diabetes Care. 2002 Nov;25(11):1952-7. doi: 10.2337/diacare.25.11.1952. PMID 12401738
- [Background] Lassmann-Vague V, Guerci B, Hanaire-Broutin H, Pinget M, Renard E, Selam JL, Vague P. Use of implantable insulin pumps: the EVADIAC position. Recommendations of ALFEDIAM (French Language Association for the Study of Diabetes and Metabolic Diseases). Evaluation dans le Diabete du Traitement par Implants Actifs. Diabetes Metab. 1997 Jun;23(3):234-50. No abstract available. English, French. PMID 9234003
- [Background] Cho JH, Chang SA, Kwon HS, Choi YH, Ko SH, Moon SD, Yoo SJ, Song KH, Son HS, Kim HS, Lee WC, Cha BY, Son HY, Yoon KH. Long-term effect of the Internet-based glucose monitoring system on HbA1c reduction and glucose stability: a 30-month follow-up study for diabetes management with a ubiquitous medical care system. Diabetes Care. 2006 Dec;29(12):2625-31. doi: 10.2337/dc05-2371. PMID 17130195
- [Background] Gold MR, Siegel JE, Russel LB, Weinstein MC. Cost-effectiveness in health and medicine. New-york : Oxford University Press, 1996.
- [Background] Frison L, Pocock SJ. Repeated measures in clinical trials: analysis using mean summary statistics and its implications for design. Stat Med. 1992 Sep 30;11(13):1685-704. doi: 10.1002/sim.4780111304. PMID 1485053
- [Background] Farmer AJ, Prevost AT, Hardeman W, Craven A, Sutton S, Griffin SJ, Kinmonth AL; Support and Advice for Medication Trial Group. Protocol for SAMS (Support and Advice for Medication Study): a randomised controlled trial of an intervention to support patients with type 2 diabetes with adherence to medication. BMC Fam Pract. 2008 Apr 11;9:20. doi: 10.1186/1471-2296-9-20. PMID 18405345
- [Background] Charpentier G, Benhamou PY, Dardari D, Clergeot A, Franc S, Schaepelynck-Belicar P, Catargi B, Melki V, Chaillous L, Farret A, Bosson JL, Penfornis A; TeleDiab Study Group. The Diabeo software enabling individualized insulin dose adjustments combined with telemedicine support improves HbA1c in poorly controlled type 1 diabetic patients: a 6-month, randomized, open-label, parallel-group, multicenter trial (TeleDiab 1 Study). Diabetes Care. 2011 Mar;34(3):533-9. doi: 10.2337/dc10-1259. Epub 2011 Jan 25. PMID 21266648
- [Background] Schaepelynck P, Renard E, Jeandidier N, Hanaire H, Fermon C, Rudoni S, Catargi B, Riveline JP, Guerci B, Millot L, Martin JF, Sola A; EVADIAC Group. A recent survey confirms the efficacy and the safety of implanted insulin pumps during long-term use in poorly controlled type 1 diabetes patients. Diabetes Technol Ther. 2011 Jun;13(6):657-60. doi: 10.1089/dia.2010.0209. Epub 2011 Apr 6. PMID 21470000
- [Background] Riveline JP, Schaepelynck P, Chaillous L, Renard E, Sola-Gazagnes A, Penfornis A, Tubiana-Rufi N, Sulmont V, Catargi B, Lukas C, Radermecker RP, Thivolet C, Moreau F, Benhamou PY, Guerci B, Leguerrier AM, Millot L, Sachon C, Charpentier G, Hanaire H; EVADIAC Sensor Study Group. Assessment of patient-led or physician-driven continuous glucose monitoring in patients with poorly controlled type 1 diabetes using basal-bolus insulin regimens: a 1-year multicenter study. Diabetes Care. 2012 May;35(5):965-71. doi: 10.2337/dc11-2021. Epub 2012 Mar 28. PMID 22456864
- [Background] Siddiqui O, Hung HM, O'Neill R. MMRM vs. LOCF: a comprehensive comparison based on simulation study and 25 NDA datasets. J Biopharm Stat. 2009;19(2):227-46. doi: 10.1080/10543400802609797. PMID 19212876
- [Background] Freudenheim JL, Johnson NE, Wardrop RL. Misclassification of nutrient intake of individuals and groups using one-, two-, three-, and seven-day food records. Am J Epidemiol. 1987 Oct;126(4):703-13. doi: 10.1093/oxfordjournals.aje.a114710. PMID 3631059
- [Result] Turnin MC, Gourdy P, Martini J, Buisson JC, Chauchard MC, Delaunay J, Schirr-Bonnans S, Taoui S, Poncet MF, Cosma V, Lablanche S, Coustols-Valat M, Chaillous L, Thivolet C, Sanz C, Penfornis A, Lepage B, Colineaux H, Mounie M, Costa N, Molinier L, Hanaire H; Educ@dom Study Group. Impact of a Remote Monitoring Programme Including Lifestyle Education Software in Type 2 Diabetes: Results of the Educ@dom Randomised Multicentre Study. Diabetes Ther. 2021 Jul;12(7):2059-2075. doi: 10.1007/s13300-021-01095-x. Epub 2021 Jun 23. PMID 34160791
- [Derived] Mounie M, Costa N, Gourdy P, Latorre C, Schirr-Bonnans S, Lagarrigue JM, Roussel H, Martini J, Buisson JC, Chauchard MC, Delaunay J, Taoui S, Poncet MF, Cosma V, Lablanche S, Coustols-Valat M, Chaillous L, Thivolet C, Sanz C, Penfornis A, Lepage B, Colineaux H, Hanaire H, Molinier L, Turnin MC; Educ@dom Study Group. Cost-Effectiveness Evaluation of a Remote Monitoring Programme Including Lifestyle Education Software in Type 2 Diabetes: Results of the Educ@dom Study. Diabetes Ther. 2022 Apr;13(4):693-708. doi: 10.1007/s13300-022-01207-1. Epub 2022 Feb 8. PMID 35133640
- See also: Simon P, Acker D. La place de la telemedicine dans l'organisation des soins. Rapport :2008 — http://www.sante.gouv.fr/IMG/pdf/Rapport_final_Telemedecine.pdf